CLINICAL TRIAL: NCT01295333
Title: Assessing the Impact of the Early and Systematic Hormonal Replacement After Radio-isotopic Ablation of Graves'hyperthyroïdism on Quality of Life, Efficiency and Tolerance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010-023608-28; 2010-23 (Other: AP HM)
Record Dates: First submitted 2011-01-27; First posted 2011-02-14 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Graves Disease (Basedow's Disease)
MeSH Terms: conditions — Graves Disease | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional approach (Other): conventional traitment
  Interventions: Drug: The initiation of LT4 as soon as the first biological signs of hypothyroidism.
- experimental approach (Experimental): early and systematic traitment
  Interventions: Drug: the early prophylactic introduction of low dose of LT4 (50 µg/d) at 15 days post-ablation

INTERVENTIONS:
Drug: the early prophylactic introduction of low dose of LT4 (50 µg/d) at 15 days post-ablation
  Arms: experimental approach
Drug: The initiation of LT4 as soon as the first biological signs of hypothyroidism.
  Arms: conventional approach

SUMMARY:
The aim of our study is to compare in a randomized multicentric study the early prophylactic introduction of low dose of LT4 (50 µg/d) at 15 days post-ablation (experimental arm) compared to a conventional approach based on the initiation of LT4 as soon as the first biological signs of hypothyroidism. Two hundred patients with Graves' disease with no or minimal (eyelid retraction or oculopalpebral asynergy) and non inflammatory ophthalmopathy (clinical activity score to 0) will be included in this study. The administrated iodine-131 activity will be adjusted to the weight of the thyroid gland (20 MBq/g thyroid tissue). Patients will be evaluated at 6 weeks, 3 months, 6 months and 12 months post-ablation. The primary objective will assess differences in terms of quality of life at 3 months using a specific questionnaire (ThyPRO). Secondary objectives will compare quality of life outcomes at different study visits (using ThyPRO and SF36), fatigue (MFIS) and depression (Beck), autoimmune parameters (signs of ophthalmopathy, TSH receptor antibodies assessment), efficacy and medico-economic data.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a hyperthyroïdie Basedowienne proving a treatment by iodine 131.

  * Patient without or with ophtalmopathie junior defined by a score of ophtalmopathie in 0 or in 1 and a score of clinical activity in 0 (see secondary).
  * Patient whose rate of fT4 and\or of fT3 is lower than 1,5 times the superior limit of the standards of the laboratory during the balance sheet(assessment) which precedes the treatment by iodine 131 (15j.
  * Patient whose thyroïdien volume estimated by echography is lower than 60 mL.
  * Patient whose treatment by anti-thyroïdiens of synthesis was interrupted at least 5 days before the administration of iodine 131.
  * 18 years old male or feminine Patient or more.

Exclusion Criteria:

* Patient presenting a thyroïdien nodule suspect of wickedness.

  * Patient presenting disorders not thyroïdiens known to distort the fixation of I131 (congestive heart failure of class III or IV, renal insufficiency).
  * Patient having received by intravenous way a product of hydrosoluble contrast for radiography in 4 weeks preceding the randomization, or by way intra-thécale or for cholécystographie by a product of contrast iodized in three months preceding the randomization.
  * Patient taking medicines susceptible to disrupt the function thyroïdienne or renal (renal medicines, lithium, amiodarone, in particular).
  * Patient presenting a contraindication to Levothyroxine with high dose: décompensée heart disorder, coronaropathie, shady of the unchecked rhythm.
  * pregnant or breast-feeding Women, or patient being able to have children and refusing to follow a reliable contraceptive method during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
will assess differences in terms of quality of life at 3 months using a specific questionnaire (ThyPRO). | 2 years

SECONDARY OUTCOMES:
compare quality of life outcomes at different study visits (using ThyPRO and SF36), fatigue (MFIS) and depression (Beck), autoimmune parameters (signs of ophthalmopathy, TSH receptor antibodies assessment), efficacy and medico-economic data. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France